CLINICAL TRIAL: NCT05048836
Title: Healthy Food First
Acronym: HFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Blue Cross Blue Shield of North Carolina (Unknown); UNC Health Alliance (Unknown); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 21-0992
Record Dates: First submitted 2021-08-31; First posted 2021-09-17 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Food Insecurity; Diet, Mediterranean
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Thus, the investigators propose conducting a 2x2x2 factorial design randomized trial to compare two food insecurity interventions, with or without a lifestyle support intervention that provides culturally tailored Med-style dietary pattern education, disease self-management support, and navigation to community resources for health related social needs, over 2 different time periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Food subsidy, no lifestyle support, 6 months (Experimental): Participant will receive $40 healthy food subsidy for 6 months.
  Interventions: Other: Food Subsidy, 6 months
- Food delivery, no lifestyle support, 6 months (Experimental): Participant will receive twice monthly healthy food delivery for 6 months.
  Interventions: Other: Food Delivery, 6 months
- Food subsidy, with lifestyle support, 6 months (Experimental): Participants will receive food subsidy and healthy lifestyle support for 6 months.
  Interventions: Other: Food Subsidy, 6 months; Behavioral: Lifestyle Support, 6 months
- Food delivery, with lifestyle support, 6 months (Experimental): Participants will receive twice monthly food box deliveries and lifestyle support for 6 months.
  Interventions: Behavioral: Lifestyle Support, 6 months; Other: Food Delivery, 6 months
- Food subsidy, no lifestyle support, 12 months (Experimental): Participants will receive food subsidy for 12 months.
  Interventions: Other: Food Subsidy, 12 months
- Food delivery, no lifestyle support, 12 months (Experimental): Participants will receive twice monthly food box deliveries for 12 months.
  Interventions: Other: Food Delivery, 12 months
- Food subsidy, with lifestyle support, 12 months (Experimental): Participant will receive food subsidy and lifestyle support for 12 months.
  Interventions: Other: Food Subsidy, 12 months; Behavioral: Lifestyle Support, 12 months
- Food delivery, with lifestyle support, 12 months (Experimental): Participants will receive twice monthly food box deliveries and lifestyle support for 12 months.
  Interventions: Behavioral: Lifestyle Support, 12 months; Other: Food Delivery, 12 months

INTERVENTIONS:
Other: Food Subsidy, 6 months — Food subsidy for 6 months
  Arms: Food subsidy, no lifestyle support, 6 months; Food subsidy, with lifestyle support, 6 months
Other: Food Subsidy, 12 months — Food subsidy for 12 months
  Arms: Food subsidy, no lifestyle support, 12 months; Food subsidy, with lifestyle support, 12 months
Behavioral: Lifestyle Support, 6 months — lifestyle support intervention delivered by community health workers for 6 months
  Arms: Food delivery, with lifestyle support, 6 months; Food subsidy, with lifestyle support, 6 months
Behavioral: Lifestyle Support, 12 months — lifestyle support intervention delivered by community health workers for 6 months
  Arms: Food delivery, with lifestyle support, 12 months; Food subsidy, with lifestyle support, 12 months
Other: Food Delivery, 6 months — Twice monthly delivery of healthy food for 6 months
  Arms: Food delivery, no lifestyle support, 6 months; Food delivery, with lifestyle support, 6 months
Other: Food Delivery, 12 months — Twice monthly delivery of healthy food for 12 months
  Arms: Food delivery, no lifestyle support, 12 months; Food delivery, with lifestyle support, 12 months

SUMMARY:
Socioeconomic barriers to healthy eating, particularly food insecurity, are a major reason for poor blood pressure control and hypertension complications. Healthy diet patterns have been shown to improve health. Unfortunately, food insecurity makes it difficult for individuals to maintain healthy diet patterns. This pragmatic randomized trial will compare two food insecurity interventions (a healthy food subsidy versus a delivered food box), with or without lifestyle support delivered by community health workers, for 6 versus 12 months duration. Key outcomes include blood pressure, food insecurity, and other patient reported outcomes.

DETAILED DESCRIPTION:
Socioeconomic barriers to healthy eating, particularly food insecurity ("insufficient or uncertain access to enough food for an active, healthy life") are a major reason for poor blood pressure control, and hypertension complications. Healthful dietary patterns, such as a Mediterranean (Med)-style diet, improve blood pressure control and reduce cardiovascular risk, risk for other chronic diseases, and premature mortality. However, food insecurity incentivizes individuals away from healthful diet patterns, resulting in wide disparities in diet-related diseases such as hypertension. Though two major ways to address food insecurity are commonly proposed-- providing subsidies for healthy food and home delivery of healthy food boxes--investigators do not know which will have the greater effect. Further, as these interventions cannot be provided indefinitely, investigators need to determine whether adding an intervention to support healthy lifestyle change, such as a culturally-tailored Med-style diet intervention, can lead to improved health even after provision of the food insecurity intervention ends.

Thus, the study team proposes to conduct 2x2x2 factorial design randomized trial to compare two food insecurity interventions, with or without a lifestyle support intervention that provides culturally tailored Med-style dietary pattern education, disease self-management support, and navigation to community resources for health related social needs, over 2 different time periods. To realize the vision of "food as medicine" to promote equity in clinical care, the study team has drawn on an extensive background of previously tested programs to create the novel multi-component interventions that will be tested in this trial. This novel intervention focuses on lowering blood pressure and addressing food insecurity. Specifically, participants will be separately randomized to receive 1) a food subsidy versus home delivery of a healthy food box, and 2) a structured lifestyle support intervention, delivered by community health workers and supervised by a registered dietitian versus usual care for 3) either 6 or 12 months. The proposed study will be conducted in central NC, enrolling 1400 participants with a history of hypertension and food insecurity. Six months after the end of each participant's intervention, investigators will re-assess study outcomes to evaluate for sustained effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension with systolic blood pressure > 130 mm Hg
* Report of food insecurity by 2-item 'Hunger Vital Sign'
* English or Spanish speaking
* Age ≥ 18 years
* Lives within delivery area of intervention services.

Exclusion Criteria:

* Pregnancy
* Malignancy
* Advanced kidney disease (estimated creatinine clearance < 30 mL/min assessed by Chronic Kidney Disease Epidemiology Collaboration formula)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Office-based Systolic Blood Pressure at Month 6 | 6 months
  Systolic blood pressure recorded at office-based healthcare visits
Office-based Systolic Blood Pressure at Month 12 | 12 months
  Systolic blood pressure recorded at office-based healthcare visits
Office-based Systolic Blood Pressure at Month 18 | 18 months
  Systolic blood pressure recorded at office-based healthcare visits
Office-based Diastolic Blood Pressure at Month 6 | 6 months
  Diastolic blood pressure recorded at office-based healthcare visits
Office-based Diastolic Blood Pressure at Month 12 | 12 months
  Diastolic blood pressure recorded at office-based healthcare visits
Office-based Diastolic Blood Pressure at Month 18 | 18 months
  Diastolic blood pressure recorded at office-based healthcare visits

SECONDARY OUTCOMES:
Ambulatory Systolic Blood Pressure at Month 6 | 6 months
  Systolic blood pressure recorded outside the healthcare system.
Ambulatory Systolic Blood Pressure at Month 12 | 12 months
  Systolic blood pressure recorded outside the healthcare system.
Ambulatory Systolic Blood Pressure at Month 18 | 18 months
  Systolic blood pressure recorded outside the healthcare system.
Ambulatory Diastolic Blood Pressure at Month 6 | 6 months
  Diastolic blood pressure recorded outside the healthcare system.
Ambulatory Diastolic Blood Pressure at Month 12 | 12 months
  Diastolic blood pressure recorded outside the healthcare system.
Ambulatory Diastolic Blood Pressure at Month 18 | 18 months
  Diastolic blood pressure recorded outside the healthcare system.
Combined (Office-based and Ambulatory) Systolic Blood Pressure at Month 6 | 6 months
  Systolic blood pressure recorded either inside or outside the healthcare system.
Combined (Office-based and Ambulatory) Systolic Blood Pressure at Month 12 | 12 months
  Systolic blood pressure recorded either inside or outside the healthcare system.
Combined (Office-based and Ambulatory) Systolic Blood Pressure at Month 18 | 18 months
  Systolic blood pressure recorded either inside or outside the healthcare system.
Combined (Office-based and Ambulatory) Diastolic Blood Pressure at Month 6 | 6 months
  Diastolic blood pressure recorded either inside or outside the healthcare system.
Combined (Office-based and Ambulatory) Diastolic Blood Pressure at Month 12 | 12 months
  Diastolic blood pressure recorded either inside or outside the healthcare system.
Combined (Office-based and Ambulatory) Diastolic Blood Pressure at Month 18 | 18 months
  Diastolic blood pressure recorded either inside or outside the healthcare system.
Food Insecurity Score at Month 6 | 6 months
  Food Insecurity Score. Score ranges from 0-10, with higher scores indicating greater food insecurity.
Food Insecurity Score at Month 12 | 12 months
  Food Insecurity Score. Score ranges from 0-10, with higher scores indicating greater food insecurity.
Food Insecurity Score at Month 18 | 18 months
  Food Insecurity Score. Score ranges from 0-10, with higher scores indicating greater food insecurity.
Health-Related Quality of Life Score as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS)-14 at Month 6 | 6 months
  The Patient-Reported Outcomes Measurement Information System(PROMIS)-14 includes seven health related quality of life domains (Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, and Pain), and the pain domain has two subdomains (interference and intensity). Raw scores, except pain intensity, are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. A higher PROMIS T-score implies more of the concept being measured; i.e., a higher PROMIS score on physical function indicates better functioning, whereas a higher score on depression indicates more severe depressive symptoms. Will report overall score and scores for each domain. From these data investigators will also calculate a PROMIS-Preference (PROPr score) (PROPr scores range from -0.022 (worst) to 1.0 (best)).
Health-Related Quality of Life Score as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS)-14 at Month 12 | 12 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) -14 includes seven health related quality of life domains (Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, and Pain), and the pain domain has two subdomains (interference and intensity). Raw scores, except pain intensity, are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. A higher PROMIS T-score implies more of the concept being measured; i.e., a higher PROMIS score on physical function indicates better functioning, whereas a higher score on depression indicates more severe depressive symptoms. Will report overall score and scores for each domain. From these data investigators will also calculate a PROMIS-Preference (PROPr score) (PROPr scores range from -0.022 (worst) to 1.0 (best)).
Health-Related Quality of Life Score as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS)-14 at Month 18 | 18 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS)-14 includes seven health related quality of life domains (Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, and Pain), and the pain domain has two subdomains (interference and intensity). Raw scores, except pain intensity, are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. A higher PROMIS T-score implies more of the concept being measured; i.e., a higher PROMIS score on physical function indicates better functioning, whereas a higher score on depression indicates more severe depressive symptoms. Will report overall score and scores for each domain. From these data investigators will also calculate a PROMIS-Preference (PROPr score) (PROPr scores range from -0.022 (worst) to 1.0 (best)).
Diet Quality at Month 6 | 6 months
  Diet Quality as assessed by Brief Dietary Assessment Scale. This score is comprised of 3 sections (or subscales) used to assess dietary patterns. Subscales are scored independently. The subscales are: Vegetables, Fruit, Whole Grains, and Beans subscale (range 0 - 20), Drinks, Desserts, Snacks, Eating Out, and Salt subscale (range 0- 20), and Fish, Meat, Poultry, Dairy, and Eggs subscale (range 0-10): Total score equals the sum of the 3 subscales. For subscales and total score, higher scores indicates better diet quality.
Diet Quality at Month 12 | 12 months
  Diet Quality as assessed by Brief Dietary Assessment Scale. This score is comprised of 3 sections (or subscales) used to assess dietary patterns. Subscales are scored independently. The subscales are: Vegetables, Fruit, Whole Grains, and Beans subscale (range 0 - 20), Drinks, Desserts, Snacks, Eating Out, and Salt subscale (range 0- 20), and Fish, Meat, Poultry, Dairy, and Eggs subscale (range 0-10): Total score equals the sum of the 3 subscales. For subscales and total score, higher scores indicates better diet quality.
Diet Quality at Month 18 | 18 months
  Diet Quality as assessed by Brief Dietary Assessment Scale. This score is comprised of 3 sections (or subscales) used to assess dietary patterns. Subscales are scored independently. The subscales are: Vegetables, Fruit, Whole Grains, and Beans subscale (range 0 - 20), Drinks, Desserts, Snacks, Eating Out, and Salt subscale (range 0- 20), and Fish, Meat, Poultry, Dairy, and Eggs subscale (range 0-10): Total score equals the sum of the 3 subscales. For subscales and total score, higher scores indicates better diet quality.
Food/ medication trade-offs at Month 6 | 6 months
  Single item-indicators of trading off medication for food or food for medication. An affirmative response indicates the presence of a trade-off.
Food/ medication trade-offs at Month 12 | 12 months
  Single item-indicators of trading off medication for food or food for medication. An affirmative response indicates the presence of a trade-off.
Food/ medication trade-offs Month 18 | 18 months
  Single item-indicators of trading off medication for food or food for medication. An affirmative response indicates the presence of a trade-off.
Diet self-efficacy at Month 6 | 6 months
  Diet Self-Efficacy as assessed by cardiac diet self-efficacy scale. Scores range from 16 to 80 with higher scores indicating greater self-efficacy.
Diet self-efficacy at Month 12 | 12 months
  Diet Self-Efficacy as assessed by cardiac diet self-efficacy scale. Scores range from 16 to 80 with higher scores indicating greater self-efficacy.
Diet self-efficacy at Month 18 | 18 months
  Diet Self-Efficacy as assessed by cardiac diet self-efficacy scale. Scores range from 16 to 80 with higher scores indicating greater self-efficacy.
Physical Activity Levels at Month 12 | 12 months
  Assessed by the International Physical Activity Questionnaire(Short Form). Higher scores indicate higher levels of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Darren DeWalt, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berkowitz SA, Ammerman AS, Knoepp P, Anderson RE 3rd, Taylor LH, Jedele JM, Archibald J, Xue K, Wertman E, Dellva B, Pignone K, Qaqish B, Dolor RJ, Turner S, Lumpkin JR, DeWalt DA. Food Insecurity Interventions to Improve Blood Pressure: The Healthy Food First Factorial Randomized Clinical Trial. JAMA Intern Med. 2025 Dec 1;185(12):1423-1433. doi: 10.1001/jamainternmed.2025.5287. PMID 41082188